CLINICAL TRIAL: NCT00813202
Title: An Open-label, Single Arm, Multi-centered Clinical Trial on the Hemodynamics and Safety of Nesiritide in the Treatment of Patients With Acute Decompensate Heart Failure
Brief Title: An Open-label, One-arm, Study to Evaluate the Hemodynamic Changes and Safety of Nesiritide for Acute Decompensated Heart Failure
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Xian-Janssen Pharmaceutical Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CR007573
Record Dates: First submitted 2008-12-18; First posted 2008-12-22 (Estimated); Last update posted 2014-02-28 (Estimated); Status verified 2014-02

CONDITIONS: Heart Decompensation; Congestive Heart Failure
Keywords: Nesiritide; Natrecor; Quanke; Acute Decompensated Heart Failure
MeSH Terms: conditions — Heart Failure | interventions — Natriuretic Peptide, Brain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Nesiritide (Experimental)
  Interventions: Drug: Nesiritide

INTERVENTIONS:
Drug: Nesiritide — Nesiritide 0.01 mcg/kg/min intravenous (IV) infusion (with or without 2 mcg/kg bolus) for 24 to 168 hours (hrs)

SUMMARY:
The present study was an open-label, uncontrolled, and multi-centered phase III clinical trial for evaluation of the efficacy (clinical efficacy and hemodynamics) and safety of nesiritide.

DETAILED DESCRIPTION:
This was an open-label, uncontrolled, and multi-centered phase II clinical trial for evaluation of the clinical efficacy and hemodynamics and safety of nesiritide. The study was conducted in hospital setting and all patients exhibited symptoms of acute decompensated heart failure, requiring treatment with intravenous drug administration. The total duration was 180 days, including a screening phase, an open treatment phase (24 hours in all) and a safety follow-up phase (day 30 and day 180). Screening phase: Right heart floating catheter was placed for patients with acute decompensate heart failure who met the inclusion criteria while not the exclusion criteria to measure pulmonary capillary wedge pressure. The results should be =20 mmHg. Open treatment phase: Nesiritide was administered by intravenous injection at a dose of 2 µg/kg for 60 second, followed by intravenous infusion at a dose of 0.01 µg/kg for 24 hour. All the patients were monitored for hemodynamics for 24 hour. Safety follow-up phase: On day 30, all the patients were required to return to the study center for follow-up. Information about death, severe adverse event, re-hospitalization and serum creatinine was collected. On day 180, all the patients were followed up by telephone. Information about death and severe adverse event was collected. Pulmonary capillary wedge pressure will be measured at 15 minutes, 1 hour, 3 hour and 24 hour, compared with baseline value. Nesiritide is white to off-white sterile lyophilized lump or powder, supplied in transparent 5 mL glass vials. The investigational drug was administered via infusion pump. Infusion rate was adjusted according to body weight. The drug was administered directly via venous cannula or the nearest injection port to the venous cannula for 60 second. The dosage of nesiritide was 2 µg/kg. The infusion rate of nesiritide was adjusted to 0.01 µg/kg/min (cannot exceed 0.01 µg/kg/min).

ELIGIBILITY:
Inclusion Criteria:

* Systolic blood pressure> 90 mmHg
* The subjects must present with dyspnoea at resting state or with minimum activity amount (such as standing up)
* Onset at this time was complicated with symptoms of acute decompensate heart failure, and it was serious enough to call for hospitalization and treatment with intravenous drug administration
* Acute decompensate heart failure was caused by cardiogenic factors rather than pulmonary factors (for example, it was neither cor pulmonale nor chronic heart failure complicated with pneumonia)
* The patients must have at least two of manifestations that related with this acute onset.

Exclusion Criteria:

* Patients with systolic blood pressure =90 mmHg
* patients who had been administered with intravenous nitroglycerin or other intravenous vasoactive drugs within 2 hour before administration of the investigational drug
* Patients who had known or suspected acute coronary syndrome (Myocardial infarction with or without increased ST segment, or unstable myocardial infarction) within 2 weeks before administration of the investigational drug
* Patients with cardiac shock or clinical manifestation of uncorrected hypovolemia or sodium depletion (such as clinical signs of excessive diuresis or dehydration), or clinical manifestation induced by other forbidden venous vasoactive agents
* Patients with such extremely emergent and unstable clinical conditions that not tolerant to Swan-Ganz catheter or temporal baseline evaluation
* patients with obvious cardiac valvular stenosis (subjects treated by valve-replacement can be included), hypertrophic, restrictive, or obstructive myocardial disease, primary pulmonary hypertension, or complex congenital heart disease.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2006-10; Primary Completion 2007-06 (Actual); Study Completion 2007-06 (Actual)

PRIMARY OUTCOMES:
Change in pulmonary capillary wedge pressure | Baseline, 180 days
  Pulmonary capillary wedge pressure will be measured in patients at all time points after administration of nesiritide, and the difference will be compared with baseline value (P<0.001).

SECONDARY OUTCOMES:
Change in clinical symptoms and overall clinical efficacy | Baseline, 180 days
  Nesiritide will attenuate dyspnoea. Nesiritide will also improve clinical symptoms and Nesiritide will improve overall clinical efficacy.

CONTACTS AND LOCATIONS:
Overall Officials: Xian-Janssen Pharmaceutical Ltd. Clinical Trial, Study Director — Xian-Janssen Pharmaceutical Ltd.
Locations (4):
- China (4):
  - Beijing
  - Hangzhou
  - Shanghai
  - Xi'an

REFERENCES:
- See also: An Open-label, Single Arm, Multi-centered Clinical Trial on the Hemodynamics and Safety of Nesiritide in the Treatment of Patients with Acute Decompensate Heart Failure — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_JNJ_6051&studyid=1093&filename=CR007573_CSR.pdf